CLINICAL TRIAL: NCT05161273
Title: Biomechanical (Fatigue-related) Risk Factors for the Development of Lower Extremity Overuse Injuries in Jump-landing Athletes
Brief Title: Risk Factors for Lower Extremity Overuse Injuries in Jump-landing Athletes
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B6702020000525-3
Record Dates: First submitted 2021-11-24; First posted 2021-12-17 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Landing Biomechanics; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective study, male jump-landing athletes (volleyball and basketball) will be screened pre-season and followed for one consecutive season. Pre-season screening consists of 3D biomechanical analysis of standardized (such as drop vertical jump) and sports-specific jumps (such as stop-jump) before and after a high-intensity, intermittent exercise protocol and clinical field tests (such as force measurements).

ELIGIBILITY:
Inclusion Criteria:

* volleyball and basketball players
* elite and non-elite
* male
* healthy

Exclusion Criteria:

* symptoms or complaints of lower extremity acute of overuse injuries in the past 3 months
* history or surgery of the lower extremities
* history of fractures of the lower extremities

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy jump-landing athletes
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Jump-landing biomechanics | 1 year
  Full-body (trunk, pelvis, hip, knee, ankle) jump-landing biomechanics (3D joint angles and moments) during drop vertical jumps, block jumps and spike jumps
Jump-landing biomechanics after fatigue | 1 year
  Full-body (trunk, pelvis, hip, knee, ankle) jump-landing biomechanics (3D joint angles and moments) during spike jumps during and after a fatigue protocol

SECONDARY OUTCOMES:
Clinical tests - force | 1 year
  Force measurements of the quadriceps, hamstrings and gluteal muscles by means of hand-held dynamometry
Clinical tests - mobility | 1 year
  Flexibility of the quadriceps and hamstrings muscles, and ankle dorsiflexion angle during dynamic weight-bearing lunge
Clinical tests - foot posture | 1 year
  Navicular height and position of the calcaneal bone
Clinical tests - force endurance | 1 year
  Prone bridge until fatigue
Clinical tests - endurance | 1 year
  Intermittent yo-yo test (level 1)

CONTACTS AND LOCATIONS:
Overall Officials: Roosen, Principal Investigator — University Ghent
Locations (1):
- Vakgroep Revalidatiewetenschappen, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided